CLINICAL TRIAL: NCT00995592
Title: Philani Home-based Nutrition Intervention Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Philani Child Health and Nutrition Project, Khayelitsha, Cape Town, South Africa (Unknown)
Responsible Party: Mary Jane Rotheram-Borus, UCLA - Center for Community Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Philani - original study
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Child Weight
Keywords: nutrition; child weight; undernourishment; mentor mother; South Africa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mentor mothers (Experimental): Behavioral intervention was offered through mentor mothers. Mentors were mothers in community who were selected by because they were doing well. They were trained to conduct home visits, up to 16 times over one year period, ranging from 20 minutes to 2 hours. Mentor mothers worked to improve health of mother and their child and build social support in neighborhood.
  Interventions: Behavioral: Philani nutrition intervention program (mentor mothers)
- Control (No Intervention): Control cases were visited and their infants were weighed 4 times over one year period. After one year, mothers were provided Philani nutrition intervention program.

INTERVENTIONS:
Behavioral: Philani nutrition intervention program (mentor mothers) — Behavioral intervention was offered through mentor mothers. Mentors were mothers in community who were selected by because they were doing well. They were trained to conduct home visits, up to 16 times over one year period, ranging from 20 minutes to 2 hours. Mentor mothers worked to improve health of mother and their child and build social support in neighborhood.
  Arms: Mentor mothers

SUMMARY:
Malnourished children and babies with birth weights under 2500 grams are at high risk for negative outcomes over their lifespan. Philani, a paraprofessional home-visiting program, was mounted in neighborhoods in three townships in Cape Town, South Africa, from 2002 to 2004 to improve nutritional outcomes.

One mentor mother was recruited from each of 37 neighborhoods. Mentor mothers were trained to conduct home visits to weigh children and to support mothers to problem-solve life challenges, especially around nutrition. Households were randomly assigned on a 2-to-1 ratio to the Philani program or to a standard care condition. Children were evaluated over a 1-year period.

The investigators hypothesized that children in the intervention would gain more weight than children in the control.

ELIGIBILITY:
Inclusion Criteria:

* mother or caregiver
* with child under 5 years of age and malnourished (malnourished if less than 2 standard deviations below the World Health Organization normative mean weight for the child's age

Exclusion Criteria:

* no malnourished children under care
* malnourished children not living in household

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2002-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
weight-for-age z-score | one year

SECONDARY OUTCOMES:
weight in kilograms | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Philani Child Health and Nutrition Project, Khayelitsha, Cape Town, South Africa

REFERENCES:
- [Derived] Christodoulou J, Rotheram-Borus MJ, Bradley AK, Tomlinson M. Home Visiting and Antenatal Depression Affect the Quality of Mother and Child Interactions in South Africa. J Am Acad Child Adolesc Psychiatry. 2019 Dec;58(12):1165-1174. doi: 10.1016/j.jaac.2019.03.016. Epub 2019 Mar 26. PMID 30926571